CLINICAL TRIAL: NCT06295835
Title: Clinical Evaluation of the Potassium (K) and Ionized Calcium (iCa) Tests in Capillary Specimens Using the i-STAT CG8+ Cartridge With the i-STAT 1 Analyzer
Brief Title: Method Comparison Study for Measuring Potassium (K) and Ionized Calcium (iCa) in Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Point of Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CS-2024-0001
Record Dates: First submitted 2024-02-26; First posted 2024-03-06 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Potassium (K) & Ionized Calcium (iCa) in Capillary Whole Blood

STUDY DESIGN:
Intervention Model Description: Capillary whole blood specimens will be tested in duplicate on the i-STAT 1 Analyzer with the CG8+ cartridge and a blood analyte testing comparator device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Method comparison for K and iCa Tests using capillary whole blood specimens. (Other): Compare the performance of the K and iCa Tests using the IUO i-STAT CG8+ Cartridge on the i-STAT 1 Analyzer to the performance of the K and iCa Tests on the comparator device using capillary whole blood specimens collected from two separate fingersticks.
  Interventions: Diagnostic Test: Fingerstick blood draw

INTERVENTIONS:
Diagnostic Test: Fingerstick blood draw — Capillary blood specimen collected from two separate fingersticks.

SUMMARY:
Method comparison study for Potassium (K) and ionized calcium (iCa).

DETAILED DESCRIPTION:
The objective of this study is to compare the performance of the K and iCa Tests using the IUO i-STAT CG8+ Cartridge on the i-STAT 1 Analyzer to the performance of the K and iCa Tests on the comparator device using capillary whole blood specimens. This objective will be assessed as part of a Method Comparison evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated consent form (if required by the IRB)
* ≥ 18 years of age

Exclusion Criteria:

• Prior enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Performance comparison | Up to 5 minutes
  Compare the performance of the Potassium (K) test using the IUO i-STAT CG8+ Cartridge on the i-STAT 1 Analyzer to the performance of the K test on a comparator device.
Performance comparison | Up to 5 minutes
  Compare the performance of the ionized calcium (iCa) test using the IUO i-STAT CG8+ Cartridge on the i-STAT 1 Analyzer to the performance of the iCa test on a comparator device.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Gupta, BS, MBA, Study Director — Abbott Point of Care
Locations (4):
- United States (3):
  - University of Maryland (UMD), Baltimore, Maryland
  - Penn State University Hershey Medical Center (Hershey), Hershey, Pennsylvania
  - Eastside Research Associates (ERA), Redmond, Washington
- Abbott Point of Care (APOC), Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No